CLINICAL TRIAL: NCT06434116
Title: Benefits of Immersive Virtual Reality on Dyspnoea During a Weaning Test in the Intensive Care Unit
Acronym: RVI-ERS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: APHP240431
Record Dates: First submitted 2024-05-23; First posted 2024-05-30 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2024-09

CONDITIONS: Spontaneous Breathing Trial in ICU
Keywords: Spontaneous breathing trial; dyspnea; virtual reality; anxiety
MeSH Terms: conditions — Dyspnea; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immersive virtual reality in patient with VAS dyspnea ≥ 3 (Experimental): Once included in the study, the patient will undergo a 15-minute session of mechanical ventilation followed by a 15-minute weaning trial without intervention (control period).
  A respiratory discomfort VAS is performed following the spontaneous breathing trial. If the VAS is ≥ 3 cm, the patient is randomised between the intervention group (immersive virtual reality) and the control group (standard care).
  The spontaneous breathing trial will be continued for a further 15 minutes in accordance with usual management, with one of the two interventions according to randomisation.
  Interventions: Device: Immersive virtual reality
- Control in patient with VAS dyspnea ≥ 3 (Experimental): Once included in the study, the patient will undergo a 15-minute session of mechanical ventilation followed by a 15-minute weaning trial without intervention (control period).
  A respiratory discomfort VAS is performed following the spontaneous breathing trial. If the VAS is ≥ 3 cm, the patient is randomised between the intervention group (immersive virtual reality) and the control group (standard care).
  The spontaneous breathing trial will be continued for a further 15 minutes in accordance with usual management, with one of the two interventions according to randomisation.
  Interventions: Device: Immersive virtual reality

INTERVENTIONS:
Device: Immersive virtual reality — The virtual reality headset is a device that simulates a realistic, three-dimensional environment, allowing the patient to be totally immersed, so that they feel as if they are really present in a virtual world. This environment can be combined with hypnotic verbal support.
  Virtual reality will be achieved using a virtual reality headset (GAMIDA®, Pico G2 4K, France) and audio headphones with noise reduction (Bose® Quiet Comfort 35 II, France). A tablet (Samsung® Galaxy Tab A 2019, 4G / Lenovo M8, France) equipped with Healthy Mind software will enable patients to enjoy a 360° visual and auditory 3D experience via a Bluetooth connection.

SUMMARY:
A weaning trial is a test that simulates physiological respiratory conditions after extubation in order to assess the patient's ability to breathe without the assistance of a ventilator.

This test is highly susceptible to induce dyspnea, with 62% of patients reporting a dyspnea score on VAS greater than 3.

Similarly, the prevalence of anxiety is high during weaning trials. 60% of patients treated in a respiratory weaning unit report psychological symptoms.

Dyspnea can be a traumatic experience for patients. In intensive care, up to half of patients suffer from dyspnea, which is described by patients as one of the worst memories of their stay in intensive care.

The virtual reality headset is a device that simulates a realistic, three-dimensional environment, allowing the patient to be totally immersed, so that they feel as if they are really present in a virtual world. This environment can be combined with hypnotic verbal support.

The research hypothesis is that virtual reality during a spontaneous breathing trial would relieve the respiratory discomfort induced by the weaning trial.

The secondary hypotheses are that virtual reality could reduce the anxiety associated with spontaneous breathing trials. These benefits could be associated to a reduction in ventilatory drive.

To assess dyspnea a VAS scale will be used, as the MV-RDOS scale, and the amplitude of EMG activity of inspiratory muscles.

DETAILED DESCRIPTION:
A weaning trial is a test that simulates physiological respiratory conditions after extubation in order to assess the patient's ability to breathe without the assistance of a ventilator.

This test is highly susceptible to induce dyspnea, with 62% of patients reporting a dyspnea score on VAS greater than 3.

Similarly, the prevalence of anxiety is high during weaning trials. 60% of patients treated in a respiratory weaning unit report psychological symptoms.

Dyspnea can be a traumatic experience for patients. In intensive care, up to half of patients suffer from dyspnea, which is described by patients as one of the worst memories of their stay in intensive care.

Dyspnea exposes patients to the risk of neuropsychological sequel, in particular the occurrence of post-traumatic stress.

Dyspnea is define by the ATS as "a subjective experience of breathing discomfort that consists of qualitatively distinct sensations that vary in intensity " . It represents a conscious and distressing sensation of breathing difficulty. It is characterized by its multidimensional aspect with a sensory and affective dimension.

To assess dyspnea a VAS scale will be used, the MV-RDOS scale, which is a recently developed tool for the hetero-assessment of dyspnea in intubated patients. The amplitude of EMG activity of the extradiaphragmatic inspiratory muscles is proportional to the intensity of dyspnea and reflects the intensity of ventilatory command. The activity of the parasternal and scalene muscles can be collected using surface electrodes.

The virtual reality headset is a device that simulates a realistic, three-dimensional environment, allowing the patient to be totally immersed, so that they feel as if they are really present in a virtual world. This environment can be combined with hypnotic verbal support.

Several studies have shown that medical hypnosis can improve the sensory and affective components of pain, and also appears to have a beneficial effect on the management of dyspnea and anxiety.

Numerous studies have shown that the use of virtual reality reduces the intensity of acute and chronic pain. Several studies have also shown that immersive virtual reality helps to reduce anxiety associated with medical procedures. A study has also found that the use of virtual reality in patients hospitalized with acute SARS-CoV-2 infection improves dyspnea, anxiety, well-being and fatigue.

The research hypothesis is that virtual reality during a spontaneous breathing trial would relieve the respiratory discomfort induced by the trial.

The secondary hypotheses are that virtual reality could reduce the anxiety associated with spontaneous breathing trials.

This will be an open label, monocentric, randomized controlled study in the intensive care unit of PItié-Salpêtrière hospital. Patient will be recruited if they are undergoing a spontaneous breathing trial as part of their usual care.

The main objective is to measure the effect of virtual reality during a ventilatory weaning trial in comparison with current practice on respiratory discomfort. Respiratory discomfort will be assessed using a visual analogue scale at the end of the ventilatory weaning trial.

The secondary objectives are to evaluate the effect of virtual reality on the intensity of anxiety, to evaluate the effect of virtual reality on respiratory discomfort assessed by the MV-RDOS score, to evaluate the effect of virtual reality on ventilatory drive assessed by the P 0.1 and EMG of scalene and parasternal muscle , to describe the effect of virtual reality on respiratory rate and heart rate, and to evaluate tolerance of virtual reality.

The study will be conducted as follows:

Once included in the study, the patient will undergo a 15-minute session of mechanical ventilation followed by a 15-minute weaning trial without intervention (control period).

A respiratory discomfort VAS is performed following the spontaneous breathing trial. If the VAS is ≥ 3 cm, the patient is randomised between the intervention group (immersive virtual reality) and the control group (standard care).

The spontaneous breathing trial will be continued for a further 15 minutes in accordance with usual care, with one of the two interventions according to randomisation.

Patients with a VAS <3 cm after the first weaning trial will not be randomised. In line with standard care, a second weaning test lasting a further 15 minutes will also be performed without intervention.

Throughout the study, the investigator will record clinical and functional data. EMG monitoring of the paraspinal and scalene muscles will be carried out throughout the test. Similarly, P 0.1 will be monitored at the beginning and end of the weaning test. The respiratory discomfort VAS, the MV-RDOS and the anxiety VAS will be assessed at the end of the weaning trial.

Completion of the sickness simulator questionnaire after the use of virtual reality in order to assess tolerance.

Virtual reality will be achieved using a virtual reality headset (GAMIDA®, Pico G2 4K, France) and audio headphones with noise reduction (Bose® Quiet Comfort 35 II, France). A tablet (Samsung® Galaxy Tab A 2019, 4G / Lenovo M8, France) equipped with Healthy Mind software will enable patients to enjoy a 360° visual and auditory 3D experience via a Bluetooth connection."

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Patients intubated and on mechanical ventilation for more than 24 hours
3. Patients eligible for a weaning trial (resolution of acute phase of pathology, low bronchial congestion, effective cough, SpO2 > 90% with Fio2 < 40%, PEEP < 8 cmH20, respiratory rate < 40/min, haemodynamically stable)
4. Decision by the doctor in charge to initiate a respiratory weaning trial as part of treatment
5. RASS score between -1 and +1
6. Patient able to answer questionnaires
7. Informed of the study and whose free and informed written consent has been obtained
8. Beneficiary of a social security plan (excluding AME)

Exclusion Criteria:

1. Non french speaker
2. Acute confusion or cognitive disorders
3. No reliable assessment of dyspnea
4. Acrophobia
5. Claustrophobia
6. Photophobia
7. Hearing loss
8. Visual impairment
9. Subject under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-03 (Estimated); Primary Completion 2025-10-03 (Estimated); Study Completion 2025-10-03 (Estimated)

PRIMARY OUTCOMES:
Respiratory discomfort VAS | At inclusion (day1)
  The primary endpoint is the comparison of the respiratory discomfort VAS between the intervention group (VR) and the control group (standard care) at the end of the ventilatory weaning test.
  Scale values:0-10, higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Effect of IVR on anxiety intensity at the end of the withdrawal test | At inclusion (day1)
  Comparison of the VAS anxiety at the end of the weaning trial between the VR group and the control group Scale values:0-10, higher scores mean a worse outcome.
Evaluation of the effect of virtual reality on respiratory discomfort assessed by the MV-RDOS (Mechanical Ventilation-Respiratory Distress Observation) score | At inclusion (day1)
  Comparison of the MV-RDOS scale between the VR group and the control group (Clinically important dyspenea is defined by MV-RDOS value ≥ 2.6)
Evaluation of the effect of virtual reality on respiratory drive assessed by the P 0.1, and EMG of scalene and parasternal muscle | At inclusion (day1)
  Evolution of physiological measurements (RMS of the parasternal and scalene EMG, P 0.1) between the VR group and the control group
Description of the effect of virtual reality on respiratory rate and heart rate | At inclusion (day1)
  Evolution of physiological measurements (respiratory rate, heart rate) between the VR group and the control group
Evaluation of the tolerance of virtual reality. | At inclusion (day1)
  Measurement of tolerance by the simulator sickness questionnaire in the VR group.

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients. Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal